CLINICAL TRIAL: NCT01769599
Title: Comparison of Initial Treatment in With Laser Grid in Diabetic Macular Edema to Intra Vitreal Avastin Injections
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Principal Investigator, yehudit.hackmon, Reaserch coordinator, Ziv Hospital
Other Study IDs: 0108-12-ZIV
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Diabetic Macular Edema; Diabetus Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Grid Treatment: 30 patients that were treated with laser grid treatment
- Avastin Treatment: patients that were treated with Avastin injections

SUMMARY:
there is no yet agreement about the best way to treat Diabetic Macular Edema (DME) the two options up to day are using Grid laser treatment Vs. Avastin injections or a combination of both in this study we want to compare the two attitudes.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with macular edema
* age 30 to 80 Yrs. old
* no previous ocular treatment
* patiens with macular edema that was shown by OCT or FA
* patients with at least 6 months follow-up after the last treatment

Exclusion Criteria:

* patients with other ocular disease (such as glaucoma etc.)
* patients with previous ocular surgery
* patiens with eye trauma
* patiens with macular edema not from DM

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic people that suffer from macular edema
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Macular thickness | 36 months
  by measuring the retinal thickness and comparing in both aproaches. and see if there is any difference.

CONTACTS AND LOCATIONS:
Locations (1):
- Ziv Medical Center, Safed, Israel